CLINICAL TRIAL: NCT07230457
Title: Prospective Evaluation of Plasma Mycobacterium Tuberculosis Cell-free DNA Sequencing as a Non-Invasive Alternative to Bronchoscopy for Diagnosing Pulmonary Tuberculosis
Brief Title: Plasma MTB cfDNA Before Bronchoscopy
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Ka Pang Chan, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: Plasma_MTB_cfDNA_FOB
Record Dates: First submitted 2025-09-30; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Tuberculosis Diagnosis
Keywords: Pulmonary tuberculosis; Cell-free DNA
MeSH Terms: conditions — Tuberculosis, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood obtained from patients with PTB and non-PTB will be stored for subsequent genetic sequencing techniques
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PTB: Patients with pulmonary tuberculosis
  Interventions: Diagnostic Test: Diagnostic Test: Plasma MTB cfDNA assay
- Non-PTB: Patients without pulmonary tuberculosis
  Interventions: Diagnostic Test: Diagnostic Test: Plasma MTB cfDNA assay

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Plasma MTB cfDNA assay — Quantitative measurement of MTB cfDNA level in the plasma

SUMMARY:
Tuberculosis (TB) remains a major global health challenge, affecting over 10 million people annually. Hong Kong carries an intermediate TB burden, with ~3,200 new cases reported yearly. Pulmonary TB (PTB), the most common form, presents diagnostic difficulties. Traditional methods like sputum smear and culture often fail in patients unable to produce adequate samples, necessitating bronchoscopy to collect bronchoalveolar lavage (BAL) for mycobacterial testing.

These limitations pose risks for patients and strain healthcare systems. Bronchoscopy is invasive, resource-intensive, and may delay treatment-especially for elderly patients with comorbidities. Blood-based inflammatory markers lack diagnostic specificity. A rapid, non-invasive alternative is urgently needed.

The investigators developed a plasma-based assay that detects Mycobacterium tuberculosis cell-free DNA (MTB cfDNA) in blood. This liquid biopsy leverages metagenomic sequencing and computational analysis to identify TB-specific genetic material while minimizing contamination. Preliminary data show excellent diagnostic performance, with area under the receiver operating characteristic curve values >0.94 for TB pleurisy.

The investigators propose a prospective clinical validation study comparing plasma MTB cfDNA testing to bronchoscopy with BAL culture and molecular testing. The primary aim is to demonstrate non-inferiority of plasma cfDNA within a 10% sensitivity margin. Secondary aims include assessing how clinical and radiological features affect test performance and evaluating the assay's ability to detect drug resistance mutations for personalized therapy.

Validation could transform TB diagnosis by offering a rapid, safe, and accurate blood test. Patients could avoid invasive procedures, receive faster diagnoses, and begin treatment sooner. Detecting resistance mutations directly from plasma would enable timely, targeted therapy-critical for addressing multidrug-resistant TB. This represents a paradigm shift toward precision medicine in TB care.

Tailored to Hong Kong's epidemiological context, this study addresses a key diagnostic gap. The approach has global relevance, with potential to improve clinical outcomes, reduce costs, and accelerate progress toward WHO's TB elimination goals.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains a global health challenge, particularly in East Asia. According to the Global TB Report by the World Health Organisation (WHO) in 2024, over 10 million people contracted TB in 2023, with 1.25 million deaths attributed to the disease. India, Indonesia and China bear the highest burden, while Hong Kong maintains an intermediate incidence, averaging 3,200 new cases annually.

Pulmonary tuberculosis (PTB) is the most common form of active TB disease. Diagnosis typically relies on detecting Mycobacterium tuberculosis (MTB) in the sputum via smear microscopy, culture, or polymerase chain reaction (PCR). However, sputum smear has limited sensitivity, culture requires 6-8 weeks, and sputum production is often difficult in certain patients. PTB may present with heterogeneous radiological features, sometimes mimicking malignancy, prompting bronchoscopy with bronchoalveolar lavage (BAL) in smear-negative patients. BAL fluid (BALF) is then tested via MTB culture, PCR, and cytology. Bronchoscopy, while informative, is invasive and poses risks for elderly patients or with cardiopulmonary comorbidities. Temporary interruption of oral anticoagulants, now widely prescribed, can lead to cardioembolic complications, contributing to up to 2.6% of stroke events. Delays in scheduling bronchoscopy and awaiting BALF MTB culture results further hinder timely diagnosis. Blood inflammatory markers are non-specific. These limitations underscore the need for a non-invasive, rapid, and accurate diagnostic tool for PTB.

Advances in sequencing technology offer new diagnostic possibilities. When bacteria die, their DNA fragments enter the bloodstream as cell-free (cfDNA). Detecting microbial cfDNA in plasma, combined with bioinformatics, provides a minimally invasive method to identify pathogens directly, outperforming blood culture or surrogate markers. Plasma MTB cfDNA is an emerging diagnostic tool. The IntelliGenome CRISPR-TB Blood Test can detect MTB cfDNA and its landmark study focused on paediatric and HIV-positive populations. However, its clinical application remains limited, with no validation in intermediate-burden regions like Hong Kong, where HIV prevalence is low.

The investigator has developed a novel targeted MTB cfDNA sequencing assay. The assay uses whole-genome-based sequencing to enrich the MTB cfDNA, followed by bioinformatic filtering to remove human DNA, distinguishing MTB from non-tuberculous Mycobacterium (NTM), and exclude microbial contaminants. A prospective study would be required to confirm diagnostic accuracy and clinical utility of this new sequencing assay. The investigators hypothesise that plasma targeted MTB cfDNA sequencing is non-inferior to BALF MTB culture and PCR in diagnostic smear-negative patients undergoing bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* Presence of respiratory indication requiring bronchoscopy
* Sputum AFB smear negative or unable to expectorate sputum for investigations

Exclusion Criteria:

* BALF collected but not sent for MTB PCR
* History of PTB or EPTB
* Concomitant use of at least two anti-TB medications for more than 14 consecutive days in the past 3 months
* Repeated bronchoscopy in the same subject within the study period
* Expected survival of less than 12 months from a different pathology
* Use of unregistered therapeutic agents in the 30 days before the study
* Consent not obtained from the subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clinical indications for undergoing bronchoscopy and BAL who meet the inclusion and exclusion criteria will be prospectively enrolled in consecutive sequences
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-10-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Area under ROC curve of MTB cfDNA assay | 27 months
  The area under ROC curve of MTB cfDNA assay in discriminating PTB and non-PTB in a prospective non-selective cohort of bronchoscopy procedures

SECONDARY OUTCOMES:
The effect of radiological features on the diagnostic performance (sensitivity and specificity) of the MTB cfDNA assay | 27 months
  To compare the diagnostic performance (sensitivity and specificity) of the MTB cfDNA assay in patients with different radiological features (cavitary vs non-cavitary)

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No